CLINICAL TRIAL: NCT06787690
Title: A Prospective Multicenter Single-arm Clinical Study to Investigate Clinical Outcomes When Cohealyx™ is Used for the Management of Full Thickness Wounds Post-surgical Excision
Brief Title: Multicenter Single-arm Trial to Investigate Clinical Outcomes When Cohealyx™ is Used for Full Thickness Wounds
Acronym: Cohealyx I
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Avita Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP011
Record Dates: First submitted 2025-01-08; First posted 2025-01-22 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Burn; Trauma Wound; Full Thickness Wounds; Surgical Wound
MeSH Terms: conditions — Burns; Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cohealyx (Experimental): Cohealyx application post surgical excision
  Interventions: Device: Cohealyx

INTERVENTIONS:
Device: Cohealyx — Cohealyx application, followed by autologous split-thickness skin graft

SUMMARY:
The goal of this study is to look at clinical outcomes when Cohealyx Collagen Matrix is used to treat full thickness wounds after surgical excision in patients that require a skin graft to heal their wounds. The main question it aims to answer is how long does it take for Cohealyx to support definitive closure.

DETAILED DESCRIPTION:
This is a prospective single-arm post-market multicenter study to evaluate clinical outcomes of Cohealyx when used to manage full thickness wounds post-surgical excision. A systematic literature review and meta-analysis were conducted to establish a performance goal for the primary effectiveness endpoint (time to autografting).

Patients with a full thickness wound where autografting is clinically indicated will be considered for participation in this study. Patients will undergo a staged surgical procedure for wound closure. In the first surgery, Cohealyx will be applied to the surgically excised wound bed within 5-days post-injury.

Following placement of Cohealyx, investigators will evaluate the wound every 3 days. Once Cohealyx has successfully integrated into the wound bed, as indicated by a robust vascularized tissue bed, the wound bed will be prepared and autografted per the investigative site's standard of care.

The study area will be evaluated with respect to Cohealyx integration, time to autografting, autograft take, healing, and safety-related adverse events.

Post-autografting, subjects will be followed for 6.5 months. Treatment-related and serious adverse events will be reported through the duration of the study. At all visits, subjects' study treatment areas as well as any donor sites dressed in PermeaDerm will be documented using digital photography.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all the following criteria to be eligible for participation:

1. The patient has a staged surgical procedure planned that requires autografting for treatment of a full thickness wound.
2. The patient is hospitalized within 3 days of injury.
3. The surgical excision occurs within 5 days post-injury.
4. The patient (or parent/guardian/legally authorized representative) is willing and able to comply with all study procedures and visit schedule.
5. The patient (or parent/guardian/legally authorized representative) agrees to abstain from any other treatment of the study area or enrollment in another interventional clinical trial for the duration of his/her participation in the study (26 weeks post-autografting).
6. In the opinion of the investigator, the patient (or parent/guardian/legally authorized representative) must be able to:

   1. Understand the full nature and purpose of the study, including possible risks and adverse events,
   2. Understand instructions, and
   3. Provide voluntary written informed consent

Exclusion Criteria:

Subjects who meet any of the following criteria are not eligible for participation:

1. Clinical signs of wound infection at study area.
2. The patient has a medical condition, is using medications or receiving treatments (e.g., immune deficiency) that may compromise patient safety or the trial evaluations or objectives.
3. The patient is unable to understand English or Spanish.
4. The patient has a known hypersensitivity to bovine-derived collagen, porcine, or aloe vera materials.
5. Presence of a medical condition where the patient's life expectancy is less than 1 year (e.g., malignancy).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2025-05-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Time for Cohealyx to generate tissue capable of supporting definitive closure | Up to 30 days
  Defined as the number of days from placement of Cohealyx until placement of an autologous split-thickness skin graft

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - University of South Alabama, Mobile, Alabama
  - Valleywise Health, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - Medstar Washington Hospital Center, Washington D.C., District of Columbia
  - Univ of Iowa, Iowa City, Iowa
  - The University of Kansas Health, Kansas City, Kansas
  - University of Louisville, Louisville, Kentucky
  - University Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mercy Hospital Springfield, Springfield, Missouri
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - University of Rochester, Rochester, New York
  - Akron Children's Hospital, Akron, Ohio
  - Ohio State University, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - JPS Health Network, Fort Worth, Texas
  - Texas Tech University, Lubbock, Texas
  - Chippenham Hospital, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No